CLINICAL TRIAL: NCT02018731
Title: Pilot Study to Assess the Efficacy of L-Citrulline and Metformin in Adults With Becker's Muscular Dystrophy
Brief Title: L-citrulline and Metformin in Becker's Muscular Dystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMD01
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Becker's Muscular Dystrophy (BMD)
Keywords: Becker's Muscular dystrophy; BMD; Metformin; L-citrulline
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Metformin; Citrulline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin and Metformin & L-Citrulline (Experimental): 1500 mg/d metformin for 6 weeks, followed by 1500 mg/d metformin and 15 g/d L-citrulline for 6 further weeks
  Interventions: Drug: Metformin and Metformin & L-Citrulline
- L-Citrulline and Metformin & L-Citrulline (Experimental): 15 g/d L-citrulline for 6 weeks, followed by 1500 mg/d metformin and 15 g/d L-citrulline for 6 further weeks
  Interventions: Drug: L-Citrulline and Metformin & L-Citrulline

INTERVENTIONS:
Drug: Metformin and Metformin & L-Citrulline
  Arms: Metformin and Metformin & L-Citrulline
Drug: L-Citrulline and Metformin & L-Citrulline
  Arms: L-Citrulline and Metformin & L-Citrulline

SUMMARY:
The purpose of the study is to compare the effects of L-citrulline and metformin and their combination therapy on muscle function and force in patients with Becker muscular dystrophy (BMD).

DETAILED DESCRIPTION:
This is a single center, not-randomized open study. The study medication consists of L-citrulline and metformin administered orally; 5g citrulline and 500mg metformin tablets will be given 3 times daily.

Half of the patients will be treated with metformin during the first 6 weeks of the study. The other patients will receive initially L-citrulline for 6 weeks, before all patients will be treated with the combination therapy (metformin and L-citrulline) for another 6 week period.

The study lasts 12 weeks and includes the screening visit and 3 further visits at baseline, week 6 and week 12.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Molecular or immunohistochemical diagnosis of BMD
* ambulant at the time point of screening

Exclusion Criteria:

* Participation in another therapeutic BMD study within the last 3 months
* Use of L-Arginine, L-Citrulline or Metformin within the last 3 months
* Other chronic disease or relevant limitation of renal, liver, heart function according to discretion of investigator
* known hypersensitivity to L-citrulline or metformin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Mean change of motor function measure (MFM) D1 subscore after 6 and 12 weeks | week 6 and week 12

SECONDARY OUTCOMES:
MFM total score and six minute walking distance (6MWD) | week 6 and week 12
Change of muscle fat content (MFC) (assessed by MRI) | week 6 and week 12
Change of muscle metabolism (assessed by dual energy x-ray absorptiometry (DEXA) and indirect calorimetry) | week 6 and week 12
Change of laboratory parameters (oxidative and nitrosative stress) | week 6 and week 12

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Fischer, MD, Principal Investigator — University Children's Hospital Basel
Locations (1):
- University Children's Hospital, Basel, Canton of Basel-City, Switzerland